

Title: Takecab Tablets Special Drug Use Surveillance "Maintenance therapy for reflux

esophagitis: Long-term use"

NCT Number: NCT03214081

Protocol Approve Date: 02-Jun-2017

Certain information within this protocol has been redacted (ie, specific content is

masked irreversibly from view with a black/blue bar) to protect either personally

identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

Named persons or organizations associated with the study.

Patient identifiers within the text, tables, or figures or in by-patient data listings.

Proprietary information, such as scales or coding systems, which are considered

confidential information under prior agreements with license holder.

Other information as needed to protect confidentiality of Takeda or partners,

personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable

information or company confidential information may be removed in their entirety if it

is considered that they do not add substantially to the interpretation of the data (eg,

appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version

was Japanese.

# Special Drug Use Surveillance Protocol Takecab Tablets Special Drug Use Surveillance "Maintenance therapy for reflux esophagitis: Long-term use"

**Sponsor** Takeda Pharmaceutical Company Limited

**Protocol Number** 

Version Number Version 2
Date of June 2, 2017

preparation

# Table of Contents

| 1.0 | Background | . 1 |
|---|---|---|
| 2.0 | Objectives | . 1 |
| 3.0 | Planned sample size and rationale | . ] |
| 3.1 | Planned sample size | . ] |
| 3.2 | Rationale | . 1 |
| 4.0 | Surveillance population | . ] |
| 5.0 | Dosage and administration. | .2 |
| 6.0 | Planned number of surveillance sites by specialty department | .2 |
| 7.0 | Methods | .2 |
| 7.1 | Duration of observation. | .2 |
| 7.2 | Request to and contract with medical institutions | . 2 |
| 7.3 | Patient enrollment method | .2 |
| 7.4 | Data entry to the survey form (electronic) and electronic signature | .3 |
| 7.5 | Actions taken for serious adverse events | .3 |
| 8.0 | Planned surveillance period | .3 |
| 9.0 | Surveillance items | .3 |
| 9.1 | Patient enrollment | .3 |
| 9.2 | Patient demographics information | . 4 |
| 9.3 | Treatment information | |
| 9.4 | Tests and observations | |
| 9.4 | 4.1 Endoscopy | |
| 9.4 | 1.2 Subjective symptoms (heartburn, acid reflux, heavy stomach feeling, early satiety, epigastric pa | in |
| | epigastric burning sensation, bloating, nausea/vomiting, belching, inappetence) | . 4 |
| 9.4 | 4.3 Liver function tests | . 5 |
| 9.4 | 1.4 Serum gastrin | . 5 |
| 9.4 | 1.5 Other items of observations | . 5 |
| 9.5 | Adverse events | . 5 |
| 10.0 | Analysis items and methods | . 8 |
| 10.1 | Disposition of patients | . 8 |
| 10.2 | Patient demographics | . 8 |
| 10.3 | Treatment details | . 8 |
| 10.4 | Safety data | . 8 |
| 10 | .4.1 Incidence of adverse events | . 8 |
| 10 | .4.2 Factors which may affect safety | . 8 |
| 10.5 | Efficacy data | |
| | .5.1 Endoscopic relapse rate | |
| | .5.2 Change of the severity of subjective symptoms | |
| | .5.3 Factors which may affect efficacy | |
| | Registration of surveillance information | |

| 12.0 | Administrative structure | 9 |
|---|---|---|
| 13.0 | Trustees | 9 |
| 14.0 | Other necessary items | 9 |
| 14.1 | Protocol amendments | 9 |
| 14.2 | Actions to be taken in response to detection of any issues or concerns | 10 |
| Append | lix Observation schedule | 9 |

# 1.0 Background

Administration of Takecab Tablets as maintenance therapy for reflux esophagitis with repeated recurrences or relapses is anticipated to be continued long-term in routine clinical settings. Administration of Takecab Tablets 10 or 20 mg once daily as maintenance therapy for reflux esophagitis was evaluated for up to 24 weeks in 406 patients in a Japanese phase III double-blind comparative study and up to 52 weeks in 305 patients in a Japanese phase III long-term study, and raised no particular safety issues. However, it would be meaningful to verify the safety of Takecab Tablets used in routine clinical practice and the consistency of the long-term safety profile with the known safety profile of the drug. Thus, the present special drug use surveillance has been planned.

This surveillance will be conducted in compliance with the Ministerial Ordinance on Good Post-Marketing Study Practice (GPSP) and relevant regulatory requirements.

# 2.0 Objectives

To evaluate the safety and efficacy of long-term use of Takecab Tablets as maintenance therapy for reflux esophagitis in routine clinical practice.

## 3.0 Planned sample size and rationale

## 3.1 Planned sample size

1,000 patients

### 3.2 Rationale

The target sample size is set to 1000 for collection of 12-month therapy data from 300 patients.

Based on the results from Takepron (lansoprazole) post-marketing surveillance\*, the percentage of patients given 12-month therapy is conservatively assumed to be 30%. Thus, a target sample size of 1000 would allow collection of 12-month therapy data from 300 patients. With the data collection from 300 patients, an adverse drug reaction (ADR) occurring with an incidence of 1% or more can be detected with a probability of at least 95%, which should allow determination of ADRs characteristic of long-term use of the drug.

# 4.0 Surveillance population

This surveillance will enroll patients who require maintenance therapy for reflux esophagitis with repeated recurrences and relapses\* and who do not meet the exclusion criteria specified below. The PRECAUTIONS section of the Takecab package insert should also be referenced.

\*Re-enrollment is prohibited for patients previously enrolled in this surveillance even if they receive re-administration for maintenance therapy.

<sup>\* &</sup>quot;Reflux esophagitis/maintenance therapy 3 to 6 months": 6-month therapy in 57%

<sup>&</sup>quot;Suppression of ulcer recurrence on low-dose aspirin: Long-term use": 12-month therapy in 79.1%

<sup>&</sup>quot;Suppression of ulcer recurrence on non-steroidal anti-inflammatory drugs: Long-term use": 12-month therapy in 46.1%

### Exclusion criteria

Patients who meet any of the following criteria will be excluded:

- (1) Patients diagnosed with Los Angeles classification (Hoshihara's modification) grade A to D disease, based on endoscopy at initiation of maintenance therapy with Takecab Tablets
- (2) Patients with a history of hypersensitivity to any ingredients of Takecab Tablets
- (3) Patients receiving atazanavir sulfate or rilpivirine hydrochloride

# 5.0 Dosage and administration

The usual adult dosage is 10 mg of vonoprazan administered orally once daily. If this is inadequately effective, the dosage may be increased to 20 mg orally once daily. The PRECAUTIONS section of the Takecab package insert should also be referenced.

6.0 Planned number of surveillance sites by specialty department
Approximately 300 sites, including the internal medicine (gastroenterology) department

### 7.0 Methods

7.1 Duration of observation

12 months

# 7.2 Request to and contract with medical institutions

The surveillance implementation will use a Web-based electronic data capture system (hereinafter referred to as PPD ") will explain to the potential surveillance investigator about the surveillance objectives and contents, as well as how to use celectronic signature and handling of the user ID and the password according to the "Surveillance Implementation Outline", "Celectronic Surveillance Implementation Outline", "Celectronic Surveillance Implementation Outline", "Celectronic Surveillance Implementation Outline", accepted, a written contract for the surveillance within the specified period will be made with the medical institution.

### 7.3 Patient enrollment method

Patients will be enrolled using a centralized enrollment method via prescribed Takecab Tablets on or after the first day of the contract period for the medical institution, the surveillance investigators will enter the patient information required for enrollment (see Section 9.1) and the electronic signature in within 14 days after the prescription of Takecab Tablets (with the day of prescription counted as zero and the day following prescription counted as "1 day after prescription").

# 7.4 Data entry to the survey form (electronic) and electronic signature

The surveillance investigator will enter data on patient demographics, treatment details, etc. and the electronic signature in coupling, roughly within 1 month after the end of required observations at Month 12 of Takecab therapy. If administration of this drug could not be confirmed, this fact should be entered (no other data are required).

For patients who discontinued treatment with Takecab Tablets for certain reasons during the observation period, the surveillance investigator will enter data on patient demographics, treatment details, etc. and the electronic signature in roughly within 1 month after the end of required observations. However, for patients who discontinued Takecab therapy because of onset of an adverse event (AE), even after the discontinuation of this drug, the surveillance investigator will continue observation as far as possible up to resolution or improvement of the adverse event. The surveillance investigator will then enter the observation result and the electronic signature in CCI

### 7.5 Actions taken for serious adverse events

If any serious AE occurs during the observation period, the surveillance investigator will immediately report it to an PPD . If requested by the PPD the surveillance investigator will provide detailed information separately.

# 8.0 Planned surveillance period

Surveillance period: March 2016 to August 31, 2018

Patient enrollment period: March 2016 to August 31, 2017 Note)

Note) No patient enrolment (via even if Takecab is prescribed by August 31, 2017.

If the total number of the enrolled patients in the entire surveillance reached the planned sample size before August 31, 2017, patient enrollment will be closed before the end of the patient enrollment period. If the patient enrollment period is shortened, the surveillance period will also be changed according to the shortened enrollment period.

# 9.0 Surveillance items

The surveillance investigator will enter data of the following items into surveillance schedule is shown in the Appendix.

### 9.1 Patient enrollment

# 1) Surveillance items

Date of prescription of Takecab Tablets for maintenance therapy, patient identification number, patient initials, sex, date of birth, assessment against the exclusion criteria

## 2) Time of data collection

At enrollment of the patient

# 9.2 Patient demographics information

### 1) Surveillance items

Time of initial onset of reflux esophagitis, inpatient/outpatient classification (at initiation of Takecab therapy), hypersensitive diathesis (presence or absence, and details), complication (presence or absence, and details), height, weight, presence or absence of *Helicobacter pylori* infection (at initiation of Takecab therapy), presence or absence of hiatus hernia, smoking history, drinking history, treatment (antacids) within 1 month before initiation of maintenance therapy for reflux esophagitis (presence or absence, name of drug, reason for use)

### 2) Time of data collection

At initiation of Takecab maintenance therapy

### 9.3 Treatment information

1) Surveillance items

Takecab therapy details (daily dose, therapy dates, and reason for discontinuation), concomitant drug details (presence or absence, name of drug, reason for use)

2) Time of data collection

From initiation of Takecab maintenance therapy to Month 12 (or discontinuation of the therapy)

### 9.4 Tests and observations

### 9.4.1 Endoscopy

1) Data items

Endoscopy (performed or not, date of endoscopy, and grade<sup>Note)</sup>

Note) The Los Angeles classification (Hoshihara's modification) grade of mucosal damage will be used.

# 2) Time of data collection

At time points of endoscopy from initiation of Takecab maintenance therapy to Month 12 (or discontinuation of the therapy)

- 9.4.2 Subjective symptoms (heartburn, acid reflux, heavy stomach feeling, early satiety, epigastric pain, epigastric burning sensation, bloating, nausea/vomiting, belching, inappetence)
  - 1) Data items

Subjective symptoms (presence or absence and severity)

2) Time of data collection

At medical interviews at initiation of Takecab maintenance therapy, Month 6, and Month 12 (or discontinuation of the therapy)

### 9.4.3 Liver function tests

## 1) Test parameters

Aspartate aminotransferase (AST), alanine aminotransferase (ALT),  $\gamma$ -glutamyl transpeptidase ( $\gamma$ -GTP), alkaline phosphatase (ALP), total bilirubin, lactate dehydrogenase (LDH)

# 2) Time of data collection

At the testing from initiation of Takecab maintenance therapy\* to Month 12 (or discontinuation of the therapy)

\*Within 1 month before initiation of Takecab maintenance therapy

# 9.4.4 Serum gastrin

1) Test parameter

Serum gastrin level

# 2) Time of data collection

At the testing from initiation of Takecab maintenance therapy\* to Month 12 (or discontinuation of the therapy)

\*Within 1 month before initiation of Takecab maintenance therapy

### 9.4.5 Other items of observations

## 1) Observation items

Presence or absence of pregnancy during the observation period (only in women)

Any pregnancy found during the observation period should be immediately notified to an PPD.

In response to a request by an PPD, the surveillance investigator will provide detailed information (wherever possible up to the outcome of pregnancy, such as premature delivery).

### 2) Time of data collection

From initiation of Takecab maintenance therapy to Month 12 (or discontinuation of the therapy)

# 9.5 Adverse events

### 1) Surveillance items

Presence or absence of AEs (see Table 1), AE term, date of onset, seriousness and reason for the assessment as serious (see Table 2), reason for discontinuation of Takecab, outcome assessment date, outcome, causal relationship to Takecab\* (see Table 3) If the outcome is "not resolved" or "unknown", or if the causal relationship is "unassessable", the event should be followed as far as possible.

Detailed event information should be collected as much as possible in the event of hepatic function disorder, fracture, gastrointestinal infection with *Clostridium difficile*, or neuroendocrine tumor.

\*If the causal relationship to Takecab is "Not related", the basis for the assessment should be recorded. If the causal relationship to Takecab is "Unassessable", the reason should be recorded.

Note) Special guidance about reporting of AEs:

Abnormal worsening of the target disease, e.g., outside the predictable range of the natural course of the disease, is regarded as an AE.

Serum gastrin can increase due to the pharmacological action of Takecab. However, if Takecab therapy is discontinued because of increased serum gastrin, this event should be handled as an AE.

## 2) Time of data collection

From initiation of Takecab maintenance therapy to Month 12 (or discontinuation of the therapy)

### Table 1 Definition of an Adverse Event

An adverse event (AE) is defined as any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product.

Note that the following events will also be handled as adverse events:

- Any manifestation in an infant breastfed by a mother taking this drug
- Any untoward manifestation in a child given this drug
- Any manifestation due to occupational exposure to this drug
- Any manifestation due to a counterfeit product of a prescription drug marketed by Takeda
- Any untoward manifestation in a patient given this drug revealed by a lawsuit or any other legal action

### **Table 2** Criteria for Serious Adverse Events

An adverse event is assessed as "serious" if it results in any of the following outcomes:

- 1. results in death (Death),
- 2. is life-threatening (Life-threatening),
- 3. requires hospitalization or prolongation of existing hospitalization (Hospitalization/Prolongation of hospitalization),
- 4. results in persistent or significant disability/incapacity (Disability),
- 5. leads to a congenital anomaly or birth defect (Congenital anomaly), or
- 6. is any other important medical event that does not fulfil 1 to 5 above.

Serious adverse events include events described in the "Takeda Medically Significant AE List".

### Takeda Medically Significant AE List

- Acute respiratory failure /Acute respiratory distress syndrome (ARDS)
- Anaphylactic shock
- Torsade de pointes / Ventricular fibrillation /
- Acute renal failure

- Ventricular tachycardia
   Malignant hypertension
- Pulmonary hypertension
- Convulsive seizure (including convulsion
- Pulmonary fibrosis (including interstitial
- and epilepsy)
- pneumonia)

- Agranulocytosis

- Neuroleptic malignant syndrome/ Malignant
- hyperthermia

- Aplastic anaemia

- Spontaneous abortion / Stillbirth and fetal death
- Toxic epidermal necrolysis /

(Stevens-Johnson syndrome)

- Confirmed or suspected transmission of infectious
- Oculomucocutaneous syndrome
- agent by a medicinal product

- Hepatic necrosis

- Confirmed or suspected endotoxin shock

- Acute hepatic failure

Table 3 Assessment of the causal relationship between an adverse event and Takecab

| Causality classification | assification Definition |
|---|---|
| Related An adverse event that follows a temporal sequence administration of this drug (including the course after withdressed of the drug), or for which possible involvement of this drug can considered, although factors other than this drug, such as primary disease, complication, concomitant drugs or concurrent treatments, may also be responsible. | |
| Not related | An adverse event that does not follow a temporal sequence from administration of this drug or that can reasonably be explained by other factors, such as the primary disease, complication, concomitant drugs or concurrent treatments. |
| Unassessable | The causality cannot be assessed because of insufficiency of |

| required information, such as temporal sequence of the event onset | | | | | |
|---|---|---|---|---|---|
| relative to administration of this drug (including the course after | | | | | |
| withdrawal of | the | drug), | primary | disease, | complication, |
| concomitant dru | concomitant drugs, and concurrent treatments. | | | | |

## 10.0 Analysis items and methods

# 10.1 Disposition of patients

Number of patients enrolled, number of patients with collected survey forms (electronic), numbers of patients for safety and efficacy analyses, number of patients excluded from analysis, reason for exclusion, etc. will be summarized.

# 10.2 Patient demographics

Patient demographic data such as sex, age, hypersensitive diathesis, and complication will be summarized.

### 10.3 Treatment details

Detailed use of Takecab and concomitant drugs will be summarized.

# 10.4 Safety data

The following data will be summarized using the safety analysis set. AEs will be coded using the MedDRA/J, and summarized by Preferred Term (PT) and System Organ Class (SOC).

# 10.4.1 Incidence of adverse events

AEs occurring during the observation period will be summarized using frequency count by event type, time of onset, seriousness, causal relationship to Takecab, etc.

### 10.4.2 Factors which may affect safety

ADRs occurring during the observation period will be summarized using frequency count, with stratification of patients according to patient demographic factors (e.g., sex, age, any renal impairment, any hepatic impairment) and treatment details (e.g., detailed use of Takecab, detailed use of concomitant drugs).

# 10.5 Efficacy data

The following data will be summarized using the efficacy analysis set.

### 10.5.1 Endoscopic relapse rate

The endoscopic relapse rate (i.e., the percentage of patients assessed as having Los Angeles classification grade A to D disease) will be calculated among patients with recorded endoscopic findings at initiation of Takecab maintenance therapy, during the therapy, and at Month 12 (or discontinuation of the therapy).

## 10.5.2 Change of the severity of subjective symptoms

The change of the severity of subjective symptoms will be summarized among patients with recorded severity of subjective symptoms at initiation of Takecab maintenance therapy and at each time point of observation after administration.

# 10.5.3 Factors which may affect efficacy

The endoscopic relapse rate will be summarized with stratification of patients according to patient demographic factors (e.g., sex, age, complication) and treatment details (e.g., detailed use of Takecab, detailed use of concomitant drugs).

# 11.0 Registration of surveillance information

Before initiation of the surveillance, Takeda Pharmaceutical Company Limited will register the surveillance information with an online public clinical trials registry:

- Japan Pharmaceutical Information Center (JAPIC) Clinical Trials Information: Japan Pharmaceutical Information Center-Clinical Trials Information

### 12.0 Administrative structure

Responsible Manager

Post-marketing surveillance manager, Takeda Pharmaceutical Company Limited

| Trustees |
|----------|
| PPD |

## 14.0 Other necessary items

# 14.1 Protocol amendments

During the surveillance period, monitoring will be performed regarding the progress of the

surveillance, occurrence of ADRs unexpected from the PRECAUTIONS and serious ADRs, any increase in the incidence of particular ADRs, validity of the surveillance items, etc., and the protocol will be reviewed and amended as necessary. If any partial change to the DOSAGE AND ADMINISTRATION, INDICATIONS, etc. is approved during the surveillance period, whether or not the protocol should be amended will be examined, and the protocol will be amended as necessary.

14.2 Actions to be taken in response to detection of any issues or concerns Whenever an issue is found regarding the safety or efficacy, the data will be investigated in detail, and necessary actions will be determined.

Appendix Observation schedule

| Time of data collection/entry | | Observation period | | | | |
|---|---|---|---|---|---|---|
| Surveillance items | | At<br>enrollmen<br>t | Start of<br>Takecab<br>maintenan<br>ce therapy | Month 6 | Month 12 | Discontin<br>uation of<br>Takecab<br>maintenan<br>ce therapy |
| | Date of prescription of Takecab | 0 | | | | |
| | Tablets for maintenance therapy | 0 | | | | |
| meni | Patient identification number | 0 | | | | |
| roll | Patient initials | 0 | | | | |
| nt er | Sex | 0 | | | | |
| Patient enrollment | Date of birth | 0 | | | | |
| | Assessment against exclusion | | | | | |
| | criteria | 0 | | | | |
| | Time of initial onset of reflux | | _ | | | |
| | esophagitis | | 0 | | | |
| | Inpatient/outpatient classification | | 0 | | | |
| | Hypersensitive diathesis | | 0 | | | |
| Patient demographics | Complication | | 0 | | | |
| grap | Height, weight | | 0 | | | |
| emo | H. pylori infection | | 0 | | | |
| ent d | Hiatus hernia | | 0 | | | |
| Patie | Smoking history | | 0 | | | |
| | Drinking history | | 0 | | | |
| | Treatment (antacids) within 1 | | | | | |
| | month of maintenance therapy | | 0 | | | |
| | for reflux esophagitis | | | | | |
| lent<br>Is | Detailed use of Takecab | | - | <u> </u> | <b></b> | 0 |
| Treatment | Detailed use of concomitant drugs | | <b>4</b> | — o — | - | 0 |
| | Endoscopy | | 4 | <u> </u> | <b>—</b> | 0 |
| ts | Subjective symptoms | | 0 | 0 | 0 | 0 |
| Assessments | Liver function tests | | <b>-</b> | ONote) | <b>-</b> | 0 |
| sess | Serum gastrin | | - | O <sup>Note)</sup> | - | 0 |
| As | Pregnancy (women only) | | 4 | — o — | <b>—</b> | 0 |
| | AE monitoring | | 4 | <u> </u> | <b></b> | 0 |
| | AE monitoring | | • | _ 0 _ | $\longrightarrow$ | 0 |

o : Performed

 $\leftarrow$   $\circ$   $\rightarrow$ Performed throughout the period

Note) From ≤1 month before initiation of Takecab maintenance therapy to Month 12

# Special Drug Use Surveillance Protocol Takecab Tablets Special Drug Use Surveillance "Maintenance therapy for reflux esophagitis: Long-term use"

**Sponsor** Takeda Pharmaceutical Company Limited

Protocol Number Vonoprazan-5003

Version Number Version 1

Date of January 7, 2016

preparation

# Table of Contents

| 1.0 | Background | . 1 |
|---|---|---|
| 2.0 | Objectives | . 1 |
| 3.0 | Planned sample size and rationale | . 1 |
| 3.1 | Planned sample size | . 1 |
| 3.2 | Rationale | . 1 |
| 4.0 | Surveillance population | . 1 |
| 5.0 | Dosage and administration. | .2 |
| 6.0 | Planned number of surveillance sites by specialty department | .2 |
| 7.0 | Methods | .2 |
| 7.1 | Duration of observation. | .2 |
| 7.2 | Request to and contract with medical institutions | . 2 |
| 7.3 | Patient enrollment method | .2 |
| 7.4 | Data entry to the survey form (electronic) and electronic signature | .3 |
| 7.5 | Actions taken for serious adverse events | .3 |
| 8.0 | Planned surveillance period | .3 |
| 9.0 | Surveillance items | .3 |
| 9.1 | Patient enrollment | . 3 |
| 9.2 | Patient demographics information | ۷. |
| 9.3 | Treatment information | . 4 |
| 9.4 | Tests and observations | . 4 |
| 9.4 | 4.1 Endoscopy | . 4 |
| 9.4 | 1.2 Subjective symptoms (heartburn, acid reflux, heavy stomach feeling, early satiety, epigastric par | in |
| | epigastric burning sensation, bloating, nausea/vomiting, belching, inappetence) | . 4 |
| 9.4 | 4.3 Liver function tests | . 5 |
| 9.4 | 1.4 Serum gastrin | . 5 |
| 9.4 | 4.5 Other items of observations | . 5 |
| 9.5 | Adverse events | . 5 |
| 10.0 | Analysis items and methods | .8 |
| 10.1 | Disposition of patients | . 8 |
| 10.2 | Patient demographics | . 8 |
| 10.3 | Treatment details | . 8 |
| 10.4 | Safety data | . 8 |
| 10 | .4.1 Incidence of adverse events | . 8 |
| 10 | .4.2 Factors which may affect safety | . 8 |
| 10.5 | Efficacy data | |
| | .5.1 Endoscopic relapse rate | |
| | .5.2 Change of the severity of subjective symptoms | |
| | .5.3 Factors which may affect efficacy | |
| | Registration of surveillance information | |

| 12.0 | Administrative structure | 9 |
|---|---|---|
| 13.0 | Trustees | 9 |
| 14.0 | Other necessary items | 9 |
| 14.1 | Protocol amendments | 9 |
| 14.2 | Actions to be taken in response to detection of any issues or concerns | 10 |
| Append | lix Observation schedule | .9 |

# 1.0 Background

Administration of Takecab Tablets as maintenance therapy for reflux esophagitis with repeated recurrences or relapses is anticipated to be continued long-term in routine clinical settings. Administration of Takecab Tablets 10 or 20 mg once daily as maintenance therapy for reflux esophagitis was evaluated for up to 24 weeks in 406 patients in a Japanese phase III double-blind comparative study and up to 52 weeks in 305 patients in a Japanese phase III long-term study, and raised no particular safety issues. However, it would be meaningful to verify the safety of Takecab Tablets used in routine clinical practice and the consistency of the long-term safety profile with the known safety profile of the drug. Thus, the present special drug use surveillance has been planned.

This surveillance will be conducted in compliance with the Ministerial Ordinance on Good Post-Marketing Study Practice (GPSP) and relevant regulatory requirements.

# 2.0 Objectives

To evaluate the safety and efficacy of long-term use of Takecab Tablets as maintenance therapy for reflux esophagitis in routine clinical practice.

## 3.0 Planned sample size and rationale

## 3.1 Planned sample size

1,000 patients

### 3.2 Rationale

The target sample size is set to 1000 for collection of 12-month therapy data from 300 patients.

Based on the results from Takepron (lansoprazole) post-marketing surveillance\*, the percentage of patients given 12-month therapy is conservatively assumed to be 30%. Thus, a target sample size of 1000 would allow collection of 12-month therapy data from 300 patients. With the data collection from 300 patients, an adverse drug reaction (ADR) occurring with an incidence of 1% or more can be detected with a probability of at least 95%, which should allow determination of ADRs characteristic of long-term use of the drug.

# 4.0 Surveillance population

This surveillance will enroll patients who require maintenance therapy for reflux esophagitis with repeated recurrences and relapses\* and who do not meet the exclusion criteria specified below. The PRECAUTIONS section of the Takecab package insert should also be referenced.

\*Re-enrollment is prohibited for patients previously enrolled in this surveillance even if they receive re-administration for maintenance therapy.

<sup>\* &</sup>quot;Reflux esophagitis/maintenance therapy 3 to 6 months": 6-month therapy in 57%

<sup>&</sup>quot;Suppression of ulcer recurrence on low-dose aspirin: Long-term use": 12-month therapy in 79.1%

<sup>&</sup>quot;Suppression of ulcer recurrence on non-steroidal anti-inflammatory drugs: Long-term use": 12-month therapy in 46.1%

### Exclusion criteria

Patients who meet any of the following criteria will be excluded:

- (1) Patients diagnosed with Los Angeles classification (Hoshihara's modification) grade A to D disease, based on endoscopy at initiation of maintenance therapy with Takecab Tablets
- (2) Patients with a history of hypersensitivity to any ingredients of Takecab Tablets
- (3) Patients receiving atazanavir sulfate or rilpivirine hydrochloride

# 5.0 Dosage and administration

The usual adult dosage is 10 mg of vonoprazan administered orally once daily. If this is inadequately effective, the dosage may be increased to 20 mg orally once daily. The PRECAUTIONS section of the Takecab package insert should also be referenced.

6.0 Planned number of surveillance sites by specialty department
Approximately 300 sites, including the internal medicine (gastroenterology) department

### 7.0 Methods

7.1 Duration of observation

12 months

# 7.2 Request to and contract with medical institutions

The surveillance implementation will use a Web-based electronic data capture system (CCI). Upon request, a medical representative of PPD (hereinafter referred to as 'PPD ") will explain to the potential surveillance investigator about the surveillance objectives and contents, as well as how to use contents and enter the electronic signature and handling of the user ID and the password according to the "Surveillance Implementation Outline", 'CCI Data Entry screen images" and contents accepted, a written contract for the surveillance within the specified period will be made with the medical institution.

### 7.3 Patient enrollment method

Patients will be enrolled using a centralized enrollment method via prescribed Takecab Tablets on or after the first day of the contract period for the medical institution, the surveillance investigators will enter the patient information required for enrollment (see Section 9.1) and the electronic signature in within 14 days after the prescription of Takecab Tablets (with the day of prescription counted as zero and the day following prescription counted as "1 day after prescription").

# 7.4 Data entry to the survey form (electronic) and electronic signature

The surveillance investigator will enter data on patient demographics, treatment details, etc. and the electronic signature in coupling, roughly within 1 month after the end of the required observations at Month 12 of Takecab therapy. If administration of this drug could not be confirmed, this fact should be entered (no other data are required).

For patients who discontinued treatment with Takecab Tablets for certain reasons during the observation period, the surveillance investigator will enter data on patient demographics, treatment details, etc. and the electronic signature in roughly within 1 month after the end of required observations. However, for patients who discontinued Takecab therapy because of onset of an adverse event (AE), even after the discontinuation of this drug, the surveillance investigator will continue observation as far as possible up to resolution or improvement of the adverse event. The surveillance investigator will then enter the observation result and the electronic signature in CCI

### 7.5 Actions taken for serious adverse events

If any serious AE occurs during the observation period, the surveillance investigator will immediately report it to an PPD If requested by the PPD the surveillance investigator will provide detailed information separately.

# 8.0 Planned surveillance period

Surveillance period: March 2016 to August 31, 2018

Patient enrollment period: March 2016 to August 31, 2017 Note)

Note) No patient enrolment (via even if Takecab is prescribed by August 31, 2017.

If the total number of the enrolled patients in the entire surveillance reached the planned sample size before August 31, 2017, patient enrollment will be closed before the end of the patient enrollment period. If the patient enrollment period is shortened, the surveillance period will also be changed according to the shortened enrollment period.

# 9.0 Surveillance items

The surveillance investigator will enter data of the following items into surveillance schedule is shown in the Appendix.

### 9.1 Patient enrollment

# 1) Surveillance items

Date of prescription of Takecab Tablets for maintenance therapy, patient identification number, patient initials, sex, date of birth, assessment against the exclusion criteria

## 2) Time of data collection

At enrollment of the patient

# 9.2 Patient demographics information

### 1) Surveillance items

Time of initial onset of reflux esophagitis, inpatient/outpatient classification (at initiation of Takecab therapy), hypersensitive diathesis (presence or absence, and details), complication (presence or absence, and details), height, weight, presence or absence of *Helicobacter pylori* infection (at initiation of Takecab therapy), presence or absence of hiatus hernia, smoking history, drinking history, treatment (antacids) within 1 month before initiation of maintenance therapy for reflux esophagitis (presence or absence, name of drug, reason for use)

### 2) Time of data collection

At initiation of Takecab maintenance therapy

### 9.3 Treatment information

1) Surveillance items

Takecab therapy details (daily dose, therapy dates, and reason for discontinuation), concomitant drug details (presence or absence, name of drug, reason for use)

2) Time of data collection

From initiation of Takecab maintenance therapy to Month 12 (or discontinuation of the therapy)

### 9.4 Tests and observations

### 9.4.1 Endoscopy

1) Data items

Endoscopy (performed or not, date of endoscopy, and grade<sup>Note)</sup>

Note) The Los Angeles classification (Hoshihara's modification) grade of mucosal damage will be used.

# 2) Time of data collection

At time points of endoscopy from initiation of Takecab maintenance therapy to Month 12 (or discontinuation of the therapy)

- 9.4.2 Subjective symptoms (heartburn, acid reflux, heavy stomach feeling, early satiety, epigastric pain, epigastric burning sensation, bloating, nausea/vomiting, belching, inappetence)
  - 1) Data items

Subjective symptoms (presence or absence and severity)

2) Time of data collection

At medical interviews at initiation of Takecab maintenance therapy, Month 6, and Month 12 (or discontinuation of the therapy)

### 9.4.3 Liver function tests

# 1) Test parameters

Aspartate aminotransferase (AST), alanine aminotransferase (ALT),  $\gamma$ -glutamyl transpeptidase ( $\gamma$ -GTP), alkaline phosphatase (ALP), total bilirubin, lactate dehydrogenase (LDH)

### 2) Time of data collection

At the testing from initiation of Takecab maintenance therapy\* to Month 12 (or discontinuation of the therapy)

\*Within 1 month before initiation of Takecab maintenance therapy

# 9.4.4 Serum gastrin

1) Test parameter

Serum gastrin level

# 2) Time of data collection

At the testing from initiation of Takecab maintenance therapy\* to Month 12 (or discontinuation of the therapy)

\*Within 1 month before initiation of Takecab maintenance therapy

### 9.4.5 Other items of observations

## 1) Observation items

Presence or absence of pregnancy during the observation period (only in women)

Any pregnancy found during the observation period should be immediately notified to an PPD

In response to a request by an PPD

the surveillance investigator will provide detailed information (wherever possible up to the outcome of pregnancy, such as premature delivery).

### 2) Time of data collection

From initiation of Takecab maintenance therapy to Month 12 (or discontinuation of the therapy)

# 9.5 Adverse events

### 1) Surveillance items

Presence or absence of AEs (see Table 1), AE term, date of onset, seriousness and reason for the assessment as serious (see Table 2), reason for discontinuation of Takecab, outcome assessment date, outcome, causal relationship to Takecab\* (see Table 3) If the outcome is "not resolved" or "unknown", or if the causal relationship is "unassessable", the event should be followed as far as possible.

Detailed event information should be collected as much as possible in the event of hepatic function disorder, fracture, gastrointestinal infection with *Clostridium difficile*, or neuroendocrine tumor.

\*If the causal relationship to Takecab is "Not related", the basis for the assessment should be recorded. If the causal relationship to Takecab is "Unassessable", the reason should be recorded.

Note) Special guidance about reporting of AEs:

Abnormal worsening of the target disease, e.g., outside the predictable range of the natural course of the disease, is regarded as an AE.

Serum gastrin can increase due to the pharmacological action of Takecab. However, if Takecab therapy is discontinued because of increased serum gastrin, this event should be handled as an AE.

## 2) Time of data collection

From initiation of Takecab maintenance therapy to Month 12 (or discontinuation of the therapy)

### Table 1 Definition of an Adverse Event

An adverse event (AE) is defined as any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product.

Note that the following events will also be handled as adverse events:

- Any manifestation in an infant breastfed by a mother taking this drug
- Any untoward manifestation in a child given this drug
- Any manifestation due to occupational exposure to this drug
- Any manifestation due to a counterfeit product of a prescription drug marketed by Takeda
- Any untoward manifestation in a patient given this drug revealed by a lawsuit or any other legal action

### **Table 2** Criteria for Serious Adverse Events

An adverse event is assessed as "serious" if it results in any of the following outcomes:

- 1. results in death (Death),
- 2. is life-threatening (Life-threatening),
- 3. requires hospitalization or prolongation of existing hospitalization (Hospitalization/Prolongation of hospitalization),
- 4. results in persistent or significant disability/incapacity (Disability),
- 5. leads to a congenital anomaly or birth defect (Congenital anomaly), or
- 6. is any other important medical event that does not fulfil 1 to 5 above.

Serious adverse events include events described in the "Takeda Medically Significant AE List".

# Takeda Medically Significant AE List

- Acute respiratory failure / Acute respiratory distress syndrome (ARDS)
- Anaphylactic shock
- Torsade de pointes / Ventricular fibrillation /
- Acute renal failure

Ventricular tachycardia - Malignant hypertension

- Pulmonary hypertension
- Convulsive seizure (including convulsion
- Pulmonary fibrosis (including interstitial
- and epilepsy)
- pneumonia)

- Agranulocytosis

- Neuroleptic malignant syndrome/ Malignant
- hyperthermia

- Aplastic anaemia

- Spontaneous abortion / Stillbirth and fetal death
- Toxic epidermal necrolysis /

(Stevens-Johnson syndrome)

- Confirmed or suspected transmission of infectious
- Oculomucocutaneous syndrome
- agent by a medicinal product

- Hepatic necrosis

- Confirmed or suspected endotoxin shock

- Acute hepatic failure

### Table 3 Assessment of the causal relationship between an adverse event and Takecab

| Causality classification | eation Definition |
|---|---|
| Related | An adverse event that follows a temporal sequence from administration of this drug (including the course after withdrawal of the drug), or for which possible involvement of this drug can be considered, although factors other than this drug, such as the primary disease, complication, concomitant drugs or concurrent treatments, may also be responsible. |
| Not related | An adverse event that does not follow a temporal sequence from administration of this drug or that can reasonably be explained by other factors, such as the primary disease, complication, concomitant drugs or concurrent treatments. |
| Unassessable | The causality cannot be assessed because of insufficiency of |

| required information, such as temporal sequence of the event onset |
|---|
| relative to administration of this drug (including the course after |
| withdrawal of the drug), primary disease, complication, |
| concomitant drugs, and concurrent treatments. |

## 10.0 Analysis items and methods

# 10.1 Disposition of patients

Number of patients enrolled, number of patients with collected survey forms (electronic), numbers of patients for safety and efficacy analyses, number of patients excluded from analysis, reason for exclusion, etc. will be summarized.

# 10.2 Patient demographics

Patient demographic data such as sex, age, hypersensitive diathesis, and complication will be summarized.

### 10.3 Treatment details

Detailed use of Takecab and concomitant drugs will be summarized.

# 10.4 Safety data

The following data will be summarized using the safety analysis set. AEs will be coded using the MedDRA/J, and summarized by Preferred Term (PT) and System Organ Class (SOC).

# 10.4.1 Incidence of adverse events

AEs occurring during the observation period will be summarized using frequency count by event type, time of onset, seriousness, causal relationship to Takecab, etc.

### 10.4.2 Factors which may affect safety

ADRs occurring during the observation period will be summarized using frequency count, with stratification of patients according to patient demographic factors (e.g., sex, age, any renal impairment, any hepatic impairment) and treatment details (e.g., detailed use of Takecab, detailed use of concomitant drugs).

# 10.5 Efficacy data

The following data will be summarized using the efficacy analysis set.

### 10.5.1 Endoscopic relapse rate

The endoscopic relapse rate (i.e., the percentage of patients assessed as having Los Angeles classification grade A to D disease) will be calculated among patients with recorded endoscopic findings at initiation of Takecab maintenance therapy, during the therapy, and at Month 12 (or discontinuation of the therapy).

## 10.5.2 Change of the severity of subjective symptoms

The change of the severity of subjective symptoms will be summarized among patients with recorded severity of subjective symptoms at initiation of Takecab maintenance therapy and at each time point of observation after administration.

# 10.5.3 Factors which may affect efficacy

The endoscopic relapse rate will be summarized with stratification of patients according to patient demographic factors (e.g., sex, age, complication) and treatment details (e.g., detailed use of Takecab, detailed use of concomitant drugs).

# 11.0 Registration of surveillance information

Before initiation of the surveillance, Takeda Pharmaceutical Company Limited will register the surveillance information with an online public clinical trials registry:

- Japan Pharmaceutical Information Center (JAPIC) Clinical Trials Information: Japan Pharmaceutical Information Center-Clinical Trials Information

# 12.0 Administrative structure

Responsible Manager

Post-marketing surveillance manager, Takeda Pharmaceutical Company Limited



### 14.0 Other necessary items

## 14.1 Protocol amendments

During the surveillance period, monitoring will be performed regarding the progress of the surveillance, occurrence of ADRs unexpected from the PRECAUTIONS and serious ADRs, any increase in the incidence of particular ADRs, validity of the surveillance items, etc., and the protocol will be reviewed and amended as necessary. If any partial change to the DOSAGE AND ADMINISTRATION, INDICATIONS, etc. is approved during the surveillance period, whether or not the protocol should be amended will be examined, and the protocol will be amended as necessary.

14.2 Actions to be taken in response to detection of any issues or concerns
Whenever an issue is found regarding the safety or efficacy, the data will be investigated in detail, and necessary actions will be determined.

Appendix Observation schedule

| Time of data collection/entry Surveillance items | | Observation period | | | | |
|---|---|---|---|---|---|---|
| | | At<br>enrollment | Start of<br>Takecab<br>maintenance<br>therapy | Month 6 | Month 12 | Discontinuat<br>ion of<br>Takecab<br>maintenance<br>therapy |
| | Date of prescription of Takecab | 0 | | | | |
| l t | Tablets for maintenance therapy | | | | | |
| men | Patient identification number | 0 | | | | |
| nroll | Patient initials | 0 | | | | |
| int e | Sex | 0 | | | | |
| Patient enrollment | Date of birth | 0 | | | | |
| | Assessment against exclusion criteria | 0 | | | | |
| | Time of initial onset of reflux esophagitis | | 0 | | | |
| | Inpatient/outpatient classification | | 0 | | | |
| | Hypersensitive diathesis | | 0 | | | |
| Patient demographics | Complication | | 0 | | | |
| grap | Height, weight | | 0 | | | |
| emo | H. pylori infection | | 0 | | | |
| ent d | Hiatus hernia | | 0 | | | |
| Patie | Smoking history | | 0 | | | |
| , , | Drinking history | | 0 | | | |
| | Treatment (antacids) within 1 | | | | | |
| | month of maintenance therapy | | 0 | | | |
| | for reflux esophagitis | | | | | |
| lent<br>Is | Detailed use of Takecab | | - | <del>-</del> 0 <del></del> | | . 0 |
| Treatment | Detailed use of concomitant drugs | | 4 | <del>-</del> 0 <del>-</del> | - | 0 |
| | Endoscopy | | • | — o — | <b>•</b> | . 0 |
| ıts | Subjective symptoms | | 0 | 0 | 0 | 0 |
| Assessments | Liver function tests | | • | O <sup>Note)</sup> | <b></b> | . 0 |
| sess | Serum gastrin | | • | O <sup>Note)</sup> | <b>-</b> | . 0 |
| As | Pregnancy (women only) | | <b>4</b> | <del>-</del> 0 <del>-</del> | | 0 |
| | AE monitoring | | <b>4</b> | <b>—</b> o <b>—</b> | - | . 0 |

o : Performed

← ○ —Performed throughout the period

Note) From ≤1 month before initiation of Takecab maintenance therapy to Month 12